CLINICAL TRIAL: NCT06337097
Title: STRICT - Surveillance With TRoponin During Immune Checkpoint Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2023-1021; NCI-2024-02687 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Immune Checkpoint Therapy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Troponin Surveillance (Experimental): Participants in Group 1, will have blood tests performed prior to each immune checkpoint inhibitor infusion for 12 weeks.
  Interventions: Diagnostic Test: Troponin surveillance
- Standard of Care (Experimental): Participants in Group 2, will have standard of care testing for any heart-related side effects of immune checkpoint inhibitors.
  Interventions: Other: Standard of care

INTERVENTIONS:
Diagnostic Test: Troponin surveillance — Troponin will be monitored prior to each immune checkpoint inhibitor infusion for the first 12 weeks of therapy.
  Arms: Troponin Surveillance
Other: Standard of care — Standard of care if symptoms arise then evaluation with cardiac biomarkers and/or further cardiac testing.
  Arms: Standard of Care

SUMMARY:
To learn if monitoring blood levels of heart injury (troponin levels) in cancer participants treated with immune checkpoint inhibitors will lead to decreased heart-related side effects.

DETAILED DESCRIPTION:
Primary Objectives:

* Myocarditis CTCAE version 5.0 grade ≥ 3
* Ventricular tachycardia (≥ 30 seconds)
* Advanced atrioventricular block
* Incident heart failure event
* Cardiovascular mortality
* Non-fatal sudden cardiac arrest
* Acute coronary syndrome
* Pericarditis
* Pericardial tamponade

Secondary Objectives:

* Time from symptom onset to diagnosis of major adverse cardiovascular events
* Time from symptom onset to diagnosis of myocarditis
* Initial hospitalization duration for the adverse cardiovascular event from primary endpoint
* Peak biomarker levels including troponin T, troponin I, creatine kinase, and creatine kinase myocardial band
* Percentage of patients with negative workup for myocarditis
* Percentage of patients requiring major cardiac testing including echocardiograms, cardiac magnetic resonance imaging, and/or invasive heart catheterization
* Duration of interruption and/or discontinuation of immune checkpoint inhibitor therapy
* Cancer progression free survival
* Time to next cancer therapy

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years old
* Plan for treatment with an immune checkpoint inhibitor as standard of care even if patient is also on an additional investigational cancer therapeutic
* Willingness to provide informed consent

Exclusion Criteria:

* Troponin T not available at screening or prior to randomization
* Inability to comply with planned study procedures
* Major adverse cardiovascular event included in the primary outcome within the 30 days prior to enrollment
* Any medical condition that could interfere with, or for which the treatment might interfere with the conduct of the study or interpretation of the study results, or that would, in the opinion of the investigator, increase the risk of the participant by participating in the study
* Any factors that, in the Investigator's opinion, are likely to interfere with study procedures, such as history of noncompliance with scheduled appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Palaskas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org